CLINICAL TRIAL: NCT03841253
Title: Treatment of Vision Disturbances Due to Corneal Irregularities by Trans-epithelial Optical Phototherapeutic Keratectomy (TE-oPTK)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Vision Clinic (Other)
Collaborators: Optana GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LO007
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Corneal Astigmatism
Keywords: Trans-epithelial phototherapeutic keratectomy; PTK; TE-PTK; Corneal epithelium; Excimer laser
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: Phase 1 will be observational comparing the software predicted refractive change to the observed refractive change. Data will be collected prospectively.
  Phase 1b will be observational comparing the software predicted refractive change to the observed refractive change. Data will be collected retrospectively.
  Phase 2 will use the software predicted refractive change to plan the refractive component of the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observational Phase 1 (Other): A trans-epithelial PTK procedure will be performed using the MEL 90 excimer laser. The refractive outcome will be compared to the refractive change predicted by the EpiMaster application software. Data is collected prospectively.
  Interventions: Procedure: Trans-epithelial PTK
- Observational Phase 1b (Other): A trans-epithelial PTK procedure will be performed using the MEL 90 excimer laser. The refractive outcome will be compared to the refractive change predicted by the EpiMaster application software. Data is collected retrospectively.
  Interventions: Procedure: Trans-epithelial PTK (retrospective data collection)
- Treatment Phase 2 (Experimental): If the transition criteria are met during the observational phase, the treatment phase will be initiated. A trans-epithelial PTK procedure will be performed using the MEL 90 excimer laser, including a refractive component according to the values determined using the EpiMaster application software.
  Interventions: Procedure: EpiMaster Application Software

INTERVENTIONS:
Procedure: Trans-epithelial PTK — The MEL 90 excimer laser will be used to ablate the corneal epithelium and stroma to a pre-defined depth, using the epithelium as a natural masking agent to smooth the stromal surface.
  Arms: Observational Phase 1
Procedure: Trans-epithelial PTK (retrospective data collection) — The MEL 90 excimer laser will be used to ablate the corneal epithelium and stroma to a pre-defined depth, using the epithelium as a natural masking agent to smooth the stromal surface.
  Arms: Observational Phase 1b
Procedure: EpiMaster Application Software — The EpiMaster Application Software imports epithelial thickness data and corneal front surface topography data, and uses this to calculate the refractive change that would be induced by a trans-epithelial PTK treatment.
  Arms: Treatment Phase 2

SUMMARY:
This study sets out to evaluate the EpiMaster application software for use in predicting the refractive change induced by a trans-epithelial phototherapeutic keratectomy (TE-PTK) procedure in eyes with irregularly irregular astigmatism. If validation criteria are met during the observational phase, the software refractive prediction will be used to plan the refractive correction in TE-PTK treatments.

DETAILED DESCRIPTION:
Complications after laser eye surgery can often result in the front surface of the eye (the cornea) becoming irregular, which causes visual symptoms such as halos, glare, starbursts, double vision, and reduced contrast sensitivity. For the past 20 years, corneal irregularities have been treated using wavefront-guided ablation, topography-guided ablation or trans-epithelial phototherapeutic keratectomy (TE-PTK). Topography-guided ablation is the most effective treatment for certain types of irregularity and works by using a laser to remove tissue from the cornea in a pattern derived from a topography scan (a measurement of the shape and curvature of the front of the eye) designed to make the corneal surface more regular.

However, topography-guided ablation is less effective for other types of irregularity. In these cases, the corneal epithelium (the layer of skin on the surface of the cornea) has changed in thickness to partially hide the irregularity on the body of the cornea under the epithelium (the stroma). The epithelium does this by becoming thinner over peaks and thickening over troughs in the stroma. Therefore, the topography measurement can only detect the proportion of the irregularity that has not been hidden by the epithelium, hence reducing its effectiveness. The preferred treatment option is TE-PTK; the laser treatment is applied onto and through the epithelium, breaking through to the stroma where the epithelium is thinnest, thus removing tissue from the peaks on the stroma resulting in a more regular surface.

The main weakness of TE-PTK is that it may unpredictably change the refraction to become more short-sighted or more long-sighted or change the astigmatism. To improve this, we have developed the Epimaster software that simulates a TE-PTK treatment and predicts the change in refraction.

The aim of the study is to validate the refractive prediction produced by the Epimaster software by comparing this to the achieved result in the patients treated. The treatment received by the patient will be the same as has been used routinely for the past 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with topographic irregularly irregular astigmatism and associated quality of vision issues, where TE-PTK would be a more effective treatment than topography-guided ablation or other therapeutic treatment options.

Medically suitable for corneal laser refractive surgery.

* Calculated residual stromal thickness ≥250 µm.
* Subjects should be 21 years of age or older.
* Contact lens wearers must stop wearing their contact lenses one week per decade of wear before baseline measurements in case of hard contact lenses and one week before baseline measurements in case of soft contact lenses.
* Patient will be able to understand the patient information and willing to sign an informed consent.
* Patient will be willing to comply with all follow-up visits and the respective examinations.

Exclusion Criteria:

* Patient not being able to tolerate local or topical anesthesia
* Autoimmune diseases
* Sicca syndrome, dry eye
* Herpes viral (herpes simplex) infections
* Herpes zoster
* Diabetes
* Pregnant or nursing women (or who are planning pregnancy during the study)
* Patients with a weight of > 135 kg
* Any residual, recurrent or acute ocular disease or abnormality of the eye, e.g.
* Cataract
* Suspected glaucoma or an intraocular pressure > 21 mm of Hg
* Corneal disease
* Corneal thinning disorder, e.g. keratoconus,
* Pellucid marginal corneal degeneration
* Dystrophy of the basal membrane
* Corneal oedema
* Exudative macular degeneration
* Infection
* Any residual, recurrent, or active abnormality of the cornea to be treated, e.g.
* Existing corneal implant
* Corneal lesion
* Unstable refraction
* Connective tissue disease
* Dry eye

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The tendency of manifest sphere, cylinder and axis | 3-12 months
  The correct tendency of manifest sphere, cylinder and axis should be achieved in 90% of cases, where tendency refers to:
  1. The sign of the predicted and the post-operative sphere is equal for predicted sphere values greater than absolute value 0.50 D (confidence limit)
  2. The sign of the predicted and the post-operative cylinder is equal (same cylinder format setting like e.g. plus cylinder format) for predicted cylinder values greater than absolute value 0.50 D (confidence limit)
  3. The cylinder axis of the predicted and the post-operative cylinder do not deviate by more than ±45° for predicted cylinder values greater than absolute value 0.50 D (confidence limit)
  4. In none of the cases the prediction in sphere and cylinder is more than absolute value 2.00 D off the post-operative values.
Standard deviation of SEpostop-SEpredicted | 12 months
  Standard deviation of SEpostop-SEpredicted at each follow-up time point (represents the scatter of the refractive outcome), where SEpredicted is the refractive outcome predicted by the EpiMaster application software.

CONTACTS AND LOCATIONS:
Locations (1):
- London Vision Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared with other researchers.

REFERENCES:
- [Background] Reinstein DZ, Archer TJ, Gobbe M. Refractive and topographic errors in topography-guided ablation produced by epithelial compensation predicted by 3D Artemis VHF digital ultrasound stromal and epithelial thickness mapping. J Refract Surg. 2012 Sep;28(9):657-63. doi: 10.3928/1081597X-20120815-02. PMID 22947295
- [Background] Reinstein DZ, Archer TJ, Gobbe M. Improved effectiveness of transepithelial PTK versus topography-guided ablation for stromal irregularities masked by epithelial compensation. J Refract Surg. 2013 Aug;29(8):526-33. doi: 10.3928/1081597X-20130719-02. PMID 23909779
- [Background] Reinstein DZ, Archer TJ, Dickeson ZI, Gobbe M. Transepithelial phototherapeutic keratectomy protocol for treating irregular astigmatism based on population epithelial thickness measurements by artemis very high-frequency digital ultrasound. J Refract Surg. 2014 Jun;30(6):380-7. doi: 10.3928/1081597X-20140508-01. PMID 24972404
- [Background] Guglielmetti S, Kirton A, Reinstein DZ, Carp GI, Archer TJ. Repair of Irregularly Irregular Astigmatism by Transepithelial Phototherapeutic Keratectomy. J Refract Surg. 2017 Oct 1;33(10):714-719. doi: 10.3928/1081597X-20170721-04. PMID 28991341
- [Background] Reinstein DZ, Archer T. Combined Artemis very high-frequency digital ultrasound-assisted transepithelial phototherapeutic keratectomy and wavefront-guided treatment following multiple corneal refractive procedures. J Cataract Refract Surg. 2006 Nov;32(11):1870-6. doi: 10.1016/j.jcrs.2006.07.016. PMID 17081871